CLINICAL TRIAL: NCT05682248
Title: Science and Technology Innovation 2030
Brief Title: Study of Brain Function Evaluation and Intervention System for Acute and Prolonged Disorders of Consciousness
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Tianjin University (Other); Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021ZD0204305
Record Dates: First submitted 2022-11-13; First posted 2023-01-12 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-12

CONDITIONS: Disorder of Consciousness
Keywords: TMS; Non-invasive neuromodulation; Brain Function Test
MeSH Terms: conditions — Consciousness Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real rTMS group (Experimental): True rTMS stimulation: 10Hz, intensity: 90% RMT, duration: 10s, interval: 30s, stimulation cycle: 1 time/day, treatment duration: 10 days;
  Interventions: Device: Transcranial magnetic stimulation
- Sham rTMS group (Placebo Comparator): sham stimulation group : intensity :0; other parameters are the same as true rTMS stimulation
  Interventions: Device: Sham Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial magnetic stimulation
  Arms: Real rTMS group
Device: Sham Transcranial magnetic stimulation — Sham Transcranial magnetic stimulation
  Arms: Sham rTMS group

SUMMARY:
The research focuses on establishing a system for validating the effectiveness of key technologies for targeted combined non-invasive interventions in awakening consciousness.

DETAILED DESCRIPTION:
Analyzed the EEG activity and brain network changes before and after stimulation by TMS stimulation of key brain regions, and correlated them with brain function. To verify the "time-frequency-space" neural mechanism of consciousness.

ELIGIBILITY:
Admission criteria for patients with prolonged disorders of consciousness (Total 200) Inclusion Criteria:(1)Age 14-80 years;(2)In accordance with the diagnostic criteria of unresponsive arousal syndrome or minimally conscious state by international research;(3)Brain Trauma, stroke and hypoxic-ischemic encephalopathy lead to disturbance of consciousness;(4) right-handed；(5)The patient's family members signed the informed consent form; Exclusion Criteria:(1)The history of mental illness and a history of hearing impairment;(2)Intracranial arterial clamp, pacemaker and other metal implants; (3)During the experiment, sedatives and other drugs that affect the excitability of the cortex;(4)The presence of uncontrolled seizures or involuntary movements;

Admission criteria for patients with acute disorders of consciousness(Total 300) Inclusion Criteria:（1)Age 14-60 years;（2）Meets diagnostic criteria for coma recognized in international studies；(3)the GCS score was less than 8; (4)Brain Trauma, stroke and hypoxic-ischemic encephalopathy lead to disturbance of consciousness;(5) right-handed；(6)The patient's family members signed the informed consent form; Exclusion Criteria:(1)The history of mental illness and a history of hearing impairment;(2)Intracranial arterial clamp, pacemaker and other metal implants; (3)During the experiment, sedatives and other drugs that affect the excitability of the cortex;(4)The presence of uncontrolled seizures or involuntary movements; Admission criteria for patients with acute disorders of consciousness;(5)No spontaneous breathing;(6)Status Epilepticus;(7)Need emergency neurosurgical treatment can not cooperate with the examination;

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Coma recovery scale-revised（CRS-R） | Assessment within 24 hours before, and 1 hour after TMS treatment
  CRS-R scale includes 6 dimensions such as audiovisual, arousal level, verbal response, motor and communication, scoring 0 to 23, the higher the score the better the neurological function, and each score reflects the presence or absence of the evaluated person and the strength of consciousness
Change from the p300 in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the p300 in event related potential(ERP)
Change from resting-state in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the spectral power and coherence by in resting-state EEG
Change from TEP in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the TMS Evoked Potential(TEP)
Change from PCI in electroencephalogram | Assessment within 24 hours before, and 1 hour after TMS treatment
  Assessment the perturbational complexity index(PCI) in TMS-EEG
Change from ROI in neuroimage techniques-PET | Assessment within 24 hours before ,and 1 hour after TMS treatment
  The distribution of 18F-FDG in the brain was analyzed according to the imaging situation, and the brain regions of interest (ROI) were outlined, and the uptake of 18F-deoxyglucose (FDG) in the patients was observed according to the brain ROI.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu hospitial, capical medical university, Beijing, China

IPD SHARING:
Plan to Share IPD: No